CLINICAL TRIAL: NCT02233569
Title: COMPARISON OF TWO DIFFERENT CONCEPTS OF MESH AND FIXATION TECHNIQUE IN THE LAPAROSCOPIC OPERATIONS FOR VENTRAL AND INCISIONAL HERNIA - A RANDOMIZED CONTROLLED MONOCENTER TRIAL.
Brief Title: Comparison of Two Mesh/Fixation Concepts for Laparoscopic Ventral and Incisional Hernia Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The high recurrence rate and the findings during the reoperations were considered as serious adverse events and were the reason for study termination.
Sponsor: Polish Hernia Study Group (Other)
Responsible Party: Principal Investigator, Maciej Pawlak, MD, Polish Hernia Study Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHvsVS
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Hernia, Abdominal; Hernia,Ventral
Keywords: Laparoscopic hernia repair; Ventral hernia; Incisional hernia; IPOM
MeSH Terms: conditions — Hernia, Abdominal; Hernia, Ventral; Incisional Hernia | interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PH (Active Comparator): Intraperitoneal onlay mesh (IPOM) repair with the use of Phisiomesh implant and Securestrap fixation device.
  Interventions: Procedure: Intraperitoneal onlay mesh (IPOM) repair with the use of Phisiomesh implant and Securestrap fixation device.; Device: ETHICON PHYSIOMESH®
- VS (Active Comparator): Intraperitoneal onlay mesh (IPOM) repair with the use of Ventralight ST implant with SorbaFix fixation device.
  Interventions: Procedure: Intraperitoneal onlay mesh (IPOM) repair with the use of Ventralight ST implant with SorbaFix fixation device.; Device: Ventralight ST implant

INTERVENTIONS:
Procedure: Intraperitoneal onlay mesh (IPOM) repair with the use of Phisiomesh implant and Securestrap fixation device. — Laparoscopic intraperitoneal onlay mesh repair for abdominal wall hernia with the use of specially designed mesh and fixation device systems: Physiomesh (mesh implant) and Securestrap (fixation device)
  Other Names: ETHICON PHYSIOMESH® Flexible Composite Mesh; ETHICON SECURESTRAP® Fixation Device
  Arms: PH
Procedure: Intraperitoneal onlay mesh (IPOM) repair with the use of Ventralight ST implant with SorbaFix fixation device. — Laparoscopic intraperitoneal onlay mesh repair for abdominal wall hernia with the use of specially designed mesh and fixation device systems: Ventralight ST (mesh implant) and SofbaFix (fixation device)
  Other Names: BARD DAVOL INC.; VENTRALIGHT™ ST Mesh; Proven Sepra® Technology in a Low Profile, Lightweight Mesh; ECHO PS™ Positioning System; SORBAFIX™Absorbable Fixation System
  Arms: VS
Device: Ventralight ST implant
  Arms: VS
Device: ETHICON PHYSIOMESH®
  Arms: PH

SUMMARY:
This is a monocenter randomized controlled trial comparing two systems of mesh and fixation device for the laparoscopic ventral and incisional hernia repair with respect to pain. It has been designed as a superiority study to proof the concept of previously published mathematical model of front abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) signed by the patient or his/her legal representative
* primary or secondary ventral hernia less than 20 cm in length and less than 11 cm in width requiring elective surgical repair
* recurrence after former abdominal hernia repair WITH MESH
* recurrence after suture abdominal hernia repair CAN be included

Exclusion Criteria:

* no written informed consent
* patient under 18 years old
* emergency surgery (incarcerated hernia)
* patients with expected life time shorter than one year for example due to generalised malignancy
* BMI exceeding 40.0kg/m²
* contaminated surgical fields
* patients on immunosuppression, steroid therapy, constant pain therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pain | 7 days after the surgery
  Presence of pain 7 days after the surgery.
Pain | 3 months after the surgery
  Presence of pain 3 months after the surgery.

SECONDARY OUTCOMES:
Number of Participants with Recurrences | up to one year
  The recurrence rate in one year followup.
Number of Participants with complications. | up to one year
  The description and percentage distribution of short and long term complications following surgery.
Pain intensity | 7 days after the surgery
  Intensity of pain measured on a visual analogue scale 7 days after the surgery
Pain intensity | 30 days after the surgery
  Intensity of pain measured on a visual analogue scale 30 days after the surgery
Pain intensity | 3 months after the surgery
  Intensity of pain measured on a visual analogue scale 3 months after the surgery.
Pain intensity | 6 months after the surgery
  Intensity of pain measured on a visual analogue scale 6 months after the surgery.

OTHER OUTCOMES:
Time of the operation | intraoperative
  The duration of the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Pawlak, MD, Principal Investigator; Maciej Śmietański, PhD, Study Director
Locations (1):
- Ceynowa Hospital, Wejherowo, Pomeranian Voivodeship, Poland

REFERENCES:
- [Background] Bansal VK, Misra MC, Kumar S, Rao YK, Singhal P, Goswami A, Guleria S, Arora MK, Chabra A. A prospective randomized study comparing suture mesh fixation versus tacker mesh fixation for laparoscopic repair of incisional and ventral hernias. Surg Endosc. 2011 May;25(5):1431-8. doi: 10.1007/s00464-010-1410-6. Epub 2010 Oct 26. PMID 20976495
- [Background] Beldi G, Wagner M, Bruegger LE, Kurmann A, Candinas D. Mesh shrinkage and pain in laparoscopic ventral hernia repair: a randomized clinical trial comparing suture versus tack mesh fixation. Surg Endosc. 2011 Mar;25(3):749-55. doi: 10.1007/s00464-010-1246-0. Epub 2010 Jul 23. PMID 20652715
- [Background] Bellows CF, Berger DH. Infiltration of suture sites with local anesthesia for management of pain following laparoscopic ventral hernia repairs: a prospective randomized trial. JSLS. 2006 Jul-Sep;10(3):345-50. PMID 17212893
- [Background] Byrd JF, Agee N, Swan RZ, Lau KN, Heath JJ, Mckillop IH, Sindram D, Martinie JB, Iannitti DA. Evaluation of absorbable and permanent mesh fixation devices: adhesion formation and mechanical strength. Hernia. 2011 Oct;15(5):553-8. doi: 10.1007/s10029-011-0826-9. Epub 2011 May 19. PMID 21594698
- [Background] Carter SA, Hicks SC, Brahmbhatt R, Liang MK. Recurrence and pseudorecurrence after laparoscopic ventral hernia repair: predictors and patient-focused outcomes. Am Surg. 2014 Feb;80(2):138-48. PMID 24480213
- [Background] Chelala E, Debardemaeker Y, Elias B, Charara F, Dessily M, Alle JL. Eighty-five redo surgeries after 733 laparoscopic treatments for ventral and incisional hernia: adhesion and recurrence analysis. Hernia. 2010 Apr;14(2):123-9. doi: 10.1007/s10029-010-0637-4. Epub 2010 Feb 14. PMID 20155431
- [Background] Clarke T, Katkhouda N, Mason RJ, Cheng BC, Algra J, Olasky J, Sohn HJ, Moazzez A, Balouch M. Fibrin glue for intraperitoneal laparoscopic mesh fixation: a comparative study in a swine model. Surg Endosc. 2011 Mar;25(3):737-48. doi: 10.1007/s00464-010-1244-2. Epub 2010 Jul 31. PMID 20680350
- [Background] Deeken CR, Abdo MS, Frisella MM, Matthews BD. Physicomechanical evaluation of absorbable and nonabsorbable barrier composite meshes for laparoscopic ventral hernia repair. Surg Endosc. 2011 May;25(5):1541-52. doi: 10.1007/s00464-010-1432-0. Epub 2010 Oct 26. PMID 20976479
- [Background] Deeken CR, Matthews BD. Ventralight ST and SorbaFix versus Physiomesh and Securestrap in a porcine model. JSLS. 2013 Oct-Dec;17(4):549-59. doi: 10.4293/108680813X13693422520125. PMID 24398196
- [Background] Eriksen JR, Bech JI, Linnemann D, Rosenberg J. Laparoscopic intraperitoneal mesh fixation with fibrin sealant (Tisseel) vs. titanium tacks: a randomised controlled experimental study in pigs. Hernia. 2008 Oct;12(5):483-91. doi: 10.1007/s10029-008-0375-z. Epub 2008 May 16. PMID 18483783
- [Background] Eriksen JR, Poornoroozy P, Jorgensen LN, Jacobsen B, Friis-Andersen HU, Rosenberg J. Pain, quality of life and recovery after laparoscopic ventral hernia repair. Hernia. 2009 Feb;13(1):13-21. doi: 10.1007/s10029-008-0414-9. Epub 2008 Aug 1. PMID 18670733
- [Background] Hanna EM, Voeller GR, Roth JS, Scott JR, Gagne DH, Iannitti DA. Evaluation of ECHO PS Positioning System in a Porcine Model of Simulated Laparoscopic Ventral Hernia Repair. ISRN Surg. 2013 May 23;2013:862549. doi: 10.1155/2013/862549. Print 2013. PMID 23762628
- [Background] Liang MK, Clapp M, Li LT, Berger RL, Hicks SC, Awad S. Patient Satisfaction, chronic pain, and functional status following laparoscopic ventral hernia repair. World J Surg. 2013 Mar;37(3):530-7. doi: 10.1007/s00268-012-1873-9. PMID 23212794
- [Background] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Background] Smietanski M, Bigda J, Iwan K, Kolodziejczyk M, Krajewski J, Smietanska IA, Gumiela P, Bury K, Bielecki S, Sledzinski Z. Assessment of usefulness exhibited by different tacks in laparoscopic ventral hernia repair. Surg Endosc. 2007 Jun;21(6):925-8. doi: 10.1007/s00464-006-9055-1. Epub 2007 Jan 23. PMID 17242988
- [Background] Szymczak C, Lubowiecka I, Tomaszewska A, Smietanski M. Investigation of abdomen surface deformation due to life excitation: implications for implant selection and orientation in laparoscopic ventral hernia repair. Clin Biomech (Bristol). 2012 Feb;27(2):105-10. doi: 10.1016/j.clinbiomech.2011.08.008. Epub 2011 Sep 15. PMID 21920647
- [Background] Wassenaar E, Schoenmaeckers E, Raymakers J, van der Palen J, Rakic S. Mesh-fixation method and pain and quality of life after laparoscopic ventral or incisional hernia repair: a randomized trial of three fixation techniques. Surg Endosc. 2010 Jun;24(6):1296-302. doi: 10.1007/s00464-009-0763-1. Epub 2009 Dec 24. PMID 20033726